CLINICAL TRIAL: NCT05267522
Title: Independent Effects of High-cholesterol (High-egg) and High-saturated Fat Diets on LDL-cholesterol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Australia (Other)
Collaborators: American Egg Board (Other)
Responsible Party: Principal Investigator, Prof. Jonathan Buckley, Dean of Programs (Human Performance), University of South Australia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 204327
Record Dates: First submitted 2022-02-02; First posted 2022-03-04 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2022-03

CONDITIONS: Hypercholesterolemia; Hyperlipidemias; Physical Inactivity; Diet, Healthy
Keywords: Cholesterol; Eggs; Saturated Fat; Low density lipoprotein cholesterol; lutein; physical activity
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Counter-balanced, cross-over trial with randomization to the starting diet will be via minimization, based on the LDL-C concentration at screening and sex. Minimization will ensure balanced LDL-C and sex between the treatment groups at commencement of each of the three diets.
Who Masked: Outcomes Assessor
Masking Description: It will not be possible to blind participants to the diet being consumed, or the research dietician assisting the participants to comply with the diets. All other research staff involved in data collection will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Egg Diet (Experimental): Egg diet, contains 2 eggs per day and limits saturated fat to 6% of energy intake. Cholesterol intake is 600mg/day. Protein and carbohydrate levels will be maintained at 20% and 40% of energy intake, respectively. This diet will be followed for 5 weeks.
  Interventions: Other: Egg diet
- Egg-free Diet (Active Comparator): Egg-free diet, limits cholesterol to 300 mg/day (no eggs) with saturated fat intake at 12% of energy intake. Protein and carbohydrate levels will be maintained at 25% and 40% of energy intake, respectively. This diet will be followed for 5 weeks.
  Interventions: Other: Egg-free Diet
- Control Diet (Active Comparator): Comparator diet based on the average Australian diet, limited to 1 egg per week, with saturated fat intake at 12% of energy intake. Cholesterol intake is 600 mg/day. Protein and carbohydrate levels will be maintained at 25% and 40% of energy intake, respectively. This diet will be followed for 5 weeks.
  Interventions: Other: Control Diet

INTERVENTIONS:
Other: Egg diet — 30% fat [6% saturated fat], 20% protein, 40% carbohydrate, 600 mg cholesterol
  Other Names: High cholesterol + low saturated fat diet
  Arms: Egg Diet
Other: Egg-free Diet — 30% fat [12% saturated fat], 25% protein, 40% carbohydrate, 300 mg cholesterol
  Other Names: Low cholesterol + high saturated fat diet
  Arms: Egg-free Diet
Other: Control Diet — 30% fat [12% saturated fat], 25% protein, 40% carbohydrate, 600 mg cholesterol
  Other Names: Average Australian Diet
  Arms: Control Diet

SUMMARY:
This study will comprise a randomized controlled, counter-balanced, cross-over trial to evaluate the independent effects of a high cholesterol (high egg), low saturated fat diet and a high saturated fat, low cholesterol diet on blood lipids. Evaluations also include analysis of physical activity as there is emerging evidence that the lutein and zeaxanthin in egg yolk may increase physical activity levels by crossing the blood-brain barrier and altering neuronal function. The study will also investigate effects on a number of novel lipoprotein parameters (particle size and particle concentrations).

DETAILED DESCRIPTION:
Eggs are high in cholesterol but low in saturated fat. Data from cross-sectional, prospective, and randomized controlled trials (RCTs), suggest that egg intake does not adversely affect blood lipids or increase cardiovascular disease (CVD) risk. In fact, there is some evidence that egg consumption may reduce CVD risk. However, to date there has been no direct comparison of the effects of a high cholesterol (high egg), low saturated fat diet and a low cholesterol, high-saturated fat diet on blood lipids, and no studies have accounted for potential effects of differences in physical activity, which can also influence the blood lipid profile. Evaluations of the effect of egg consumption on blood lipids should include analysis of physical activity as there is emerging evidence that the lutein and zeaxanthin in egg yolk may increase physical activity levels by crossing the blood-brain barrier and altering neuronal function. We will directly compare the effects of a high cholesterol, low saturated fat diet and a low cholesterol, high saturated fat diet on blood lipids, using egg consumption to manipulate dietary cholesterol intake, while also accounting for physical activity levels. The study will investigate effects on a number of novel lipoprotein parameters (particle size and particle concentrations).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 - 60 years
* Blood LDL-C <3.5 mmol/L (measured at screening using an automated analyser (Cholestech LDX System).
* Non-smoker (or other nicotine products) (minimum 6 months).

Exclusion Criteria:

* Have diagnosed cardiovascular disease (including uncontrolled high blood pressure) or a chronic disease, including Type-1 or -2 diabetes, kidney or liver disease, gastrointestinal disorders requiring medical nutrition therapy (e.g., Crohn's disease, irritable bowel, coeliac disease) or any other condition that may have an impact on study outcomes.
* Have allergies or strong aversion to eggs or other components of the test foods (diets are not suitable for vegetarians).
* Consume more than 5 eggs per week in the month prior to beginning the trial.
* Participant has a recent history (within 12 months) or strong potential for alcohol abuse. Defined as >14 standard drinks per week.
* Have changed medication or supplementation that might affect study outcomes in the last 3 months.
* Take vitamin, mineral, herbal supplementation, or medications that may have an impact on study outcomes.
* Are already involved in another research project within 30 days of commencement of the present study that in the opinion of the investigators will be unsuitable for this study.
* Are pregnant or breastfeeding.
* Show unwillingness to be randomized to either experimental group.
* Failure to satisfy the investigator regarding suitability to participate for any other reason.
* Are unwilling or unable to provide written informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Low-density lipoprotein cholesterol (LDL-C) | Baseline
  Plasma LDL-C levels (mmol/L)
Low-density lipoprotein cholesterol (LDL-C) | 5 weeks
  Plasma LDL-C levels (mmol/L)
Low-density lipoprotein cholesterol (LDL-C) | 10 weeks
  Plasma LDL-C levels (mmol/L)
Low-density lipoprotein cholesterol (LDL-C) | 15 weeks
  Plasma LDL-C levels (mmol/L)

SECONDARY OUTCOMES:
Blood lipid profiling | Baseline
  Plasma lipid, lipoprotein subclasses, cholesterol, and apolipoproteins
Blood lipid profiling | 5 weeks
  Plasma lipid, lipoprotein subclasses, cholesterol, and apolipoproteins
Blood lipid profiling | 10 weeks
  Plasma lipid, lipoprotein subclasses, cholesterol, and apolipoproteins
Blood lipid profiling | 15 weeks
  Plasma lipid, lipoprotein subclasses, cholesterol, and apolipoproteins
Fasting glucose | Baseline
  Plasma glucose levels (mmol/L)
Fasting glucose | 5 weeks
  Plasma glucose levels (mmol/L)
Fasting glucose | 10 weeks
  Plasma glucose levels (mmol/L)
Fasting glucose | 15 weeks
  Plasma glucose levels (mmol/L)
Physical activity levels | Baseline
  Amount of time (min) spent sedentary and engaged in light or moderate-vigorous physical activity
Physical activity levels | 5 weeks
  Amount of time (min) spent sedentary and engaged in light or moderate-vigorous physical activity
Physical activity levels | 10 weeks
  Amount of time (min) spent sedentary and engaged in light or moderate-vigorous physical activity
Physical activity levels | 15 weeks
  Amount of time (min) spent sedentary and engaged in light or moderate-vigorous physical activity
Waist circumference | Baseline
  Waist circumference (cm) measured at the midpoint between the lower costal (10th rib) border and the iliac crest.
Waist circumference | 5 weeks
  Waist circumference (cm) measured at the midpoint between the lower costal (10th rib) border and the iliac crest.
Waist circumference | 10 weeks
  Waist circumference (cm) measured at the midpoint between the lower costal (10th rib) border and the iliac crest.
Waist circumference | 15 weeks
  Waist circumference (cm) measured at the midpoint between the lower costal (10th rib) border and the iliac crest.
Blood Pressure | Baseline
  Seated blood pressure (mmHg)
Blood Pressure | 5 weeks
  Seated blood pressure (mmHg)
Blood Pressure | 10 weeks
  Seated blood pressure (mmHg)
Blood Pressure | 15 weeks
  Seated blood pressure (mmHg)
Dietary saturated fat intake | Baseline
  Analysis of dietary intake based on 5-day food diaries
Dietary saturated fat intake | 5 weeks
  Analysis of dietary intake based on 5-day food diaries
Dietary saturated fat intake | 10 weeks
  Analysis of dietary intake based on 5-day food diaries
Dietary saturated fat intake | 15 weeks
  Analysis of dietary intake based on 5-day food diaries
Dietary cholesterol intake | Baseline
  Analysis of dietary intake based on 5-day food diaries
Dietary cholesterol intake | 5 weeks
  Analysis of dietary intake based on 5-day food diaries
Dietary cholesterol intake | 10 weeks
  Analysis of dietary intake based on 5-day food diaries
Dietary cholesterol intake | 15 weeks
  Analysis of dietary intake based on 5-day food diaries
Dietary Energy intake | Baseline
  Analysis of dietary intake based on 5-day food diaries
Dietary Energy intake | 5 weeks
  Analysis of dietary intake based on 5-day food diaries
Dietary Energy intake | 10 weeks
  Analysis of dietary intake based on 5-day food diaries
Dietary Energy intake | 15 weeks
  Analysis of dietary intake based on 5-day food diaries
Dietary Macronutrients | Baseline
  Analysis of dietary intake based on food diaries
Dietary Macronutrients | 5 weeks
  Analysis of dietary intake based on food diaries
Dietary Macronutrients | 10 weeks
  Analysis of dietary intake based on food diaries
Dietary Macronutrients | 15 weeks
  Analysis of dietary intake based on food diaries
Dietary Lutein+Zeaxanthin | Baseline
  Analysis of dietary intake based on food diaries
Dietary Lutein+Zeaxanthin | 5 weeks
  Analysis of dietary intake based on food diaries
Dietary Lutein+Zeaxanthin | 10 weeks
  Analysis of dietary intake based on food diaries
Dietary Lutein+Zeaxanthin | 15 weeks
  Analysis of dietary intake based on food diaries
Sleep | Baseline
  Sleep patterns assessed using accelerometers
Sleep | 5 weeks
  Sleep patterns assessed using accelerometers
Sleep | 10 weeks
  Sleep patterns assessed using accelerometers
Sleep | 15 weeks
  Sleep patterns assessed using accelerometers

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Buckley, PhD, Principal Investigator — University of South Australia
Locations (1):
- University of South Australia Clinical Trial Facility, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carter S, Hill AM, Yandell C, Wood L, Coates AM, Buckley JD. Impact of dietary cholesterol from eggs and saturated fat on LDL cholesterol levels: a randomized cross-over study. Am J Clin Nutr. 2025 Jul;122(1):83-91. doi: 10.1016/j.ajcnut.2025.05.001. Epub 2025 May 6. PMID 40339906
- [Derived] Carter S, Hill AM, Yandell C, Buckley JD, Coates AM. Study protocol for a 15-week randomised controlled trial assessing the independent effects of high-cholesterol and high-saturated fat diets on LDL cholesterol. BMJ Open. 2024 Jan 25;14(1):e081664. doi: 10.1136/bmjopen-2023-081664. PMID 38272555